CLINICAL TRIAL: NCT05127850
Title: Mhealth ElectroNic COnsultation REcording (MENCORE-2): an Implementation Trial to Improve Informed Treatment Decision-making in Men With Advanced Prostate Cancer
Brief Title: MENCORE-2: Audio Recordings to Improve Decision-making in Advanced Prostate Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Conquer Cancer Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 21559; NCI-2021-11595 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2021-11-08; First posted 2021-11-19 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Prostate Cancer; Metastatic Prostate Cancer; Metastatic Castration-resistant Prostate Cancer
Keywords: Consultation audio recordings; Shared decision-making
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Consultation audio recording (Experimental): Instructions on installation and detailed use of chosen application will be provided before an upcoming oncology visit. Research staff will contact the participant and encourage a "practice" recording session. 15-30 minutes prior to the consultation, research staff will send an anonymous text message to the participants' mobile device with a reminder to record the visit. Three days after the consultation, research staff will send an anonymous text reminder message to the participants' mobile device to listen to the recording.
  Interventions: Behavioral: Consultation audio recording app

INTERVENTIONS:
Behavioral: Consultation audio recording app — Smartphone or tablet mobile application which allows for voice recording
  Other Names: Voice Recording app; Mobile voice recording app; Smartphone voice recording app; Tablet voice recording app

SUMMARY:
This is a single-arm hybrid implementation trial of men with metastatic castrate-resistant prostate cancer (mCRPC) involving a patient-administered mobile app for consultation audio recordings.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

1. To evaluate change in participant informed decision-making after provision of a consultation audio recording application.

SECONDARY OBJECTIVES:

1. Reach. To evaluate the percentage of invited participants who enroll. Reasons for not enrolling will be assessed.
2. Adoption. To evaluate the percentage of providers who agree to be recorded.
3. Adoption. To evaluate the percentage of participants who create an audio recording.
4. Adoption. To evaluate the percentage of participants who listen to the audio recording or read its automatically generated transcript.
5. Implementation. To evaluate the percentage of participants who report receiving instructions on how to record.
6. To evaluate participant-reported shared decision-making effort.
7. To evaluate whether participant-reported anxiety changes after provision of a consultation audio recording app.
8. To evaluate barriers, facilitators, and experiences of recording app use, particularly in the context of treatment decision-making by conducting participant interviews, provider surveys, and interviews with providers.
9. Treatment received.

EXPLORATORY OBJECTIVES:

1. To evaluate whether provision of a consultation audio recording app improves participant-reported knowledge retention of docetaxel.
2. To evaluate accuracy of app auto-generated transcription.
3. To evaluate degree of provider decision support and communication skills.

Participants are set up with an application prior to the first physician visit and then followed-up 7 days, 28 days and 60 days after their physician encounter.

ELIGIBILITY:
Inclusion Criteria:

1. Metastatic castration-resistant prostate cancer (mCRPC) with progression per any Prostate Cancer Working Group 3 (PCWG3) criterion (Prostate-specific antigen (PSA), clinical, or radiographic)
2. Has never received any chemotherapy for prostate cancer.
3. Current or prior receipt of at least one androgen-signaling inhibitors (ASI) (abiraterone, enzalutamide, apalutamide, or darolutamide), with progression on it.
4. Eligible for docetaxel chemotherapy at any dose level (treating provider's discretion).
5. Has an upcoming genitourinary (GU) medical oncology appointment (in-person, telephone, or Zoom video visit) at University of California, San Francisco (UCSF) within 7-60 days of enrollment, during which next-line treatment options are anticipated to be discussed (treating provider's discretion).
6. 18 years of age or older.
7. Able to read, speak, and write in English (the application is in English only)
8. Has access to and ability to use an iOS or Android smartphone or tablet.
9. For video visits only: has access to and ability to use a second device (e.g., desktop, laptop, smartphone, tablet, etc.) that will run a Zoom video visit.
10. Patient's provider of the upcoming appointment in #5 agrees to be recorded.

Inclusion criteria (provider participants):

1. UCSF GU medical oncology providers (medical doctor (MD), nurse practitioner (NP), or physician's assistant (PA)), regardless of whether their patient was enrolled

Exclusion Criteria:

1. Lack of decision-making capacity to provide consent to this trial.
2. Uncorrectable hearing or visual impairment hindering the ability to perform necessary tasks in the trial.
3. Any neurocognitive or psychiatric disorder hindering the ability to perform necessary tasks in the trial.
4. Prior participation in Mobile Health ElectroNic COnsultation REcording (mENCORE) (participants have already received the intervention).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2022-03-22 (Actual); Primary Completion 2024-02-16 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Mean change in docetaxel knowledge score over time | Up to 2 weeks
  Change in docetaxel knowledge score is measured by participant report of knowledge using a docetaxel knowledge instrument, measured at baseline and 7 days post-appointment. The instrument was developed based on facts that patients and providers deem are important when making a treatment decision that includes docetaxel as an option for mCRPC (e.g., disease, prognosis, risks, benefits, alternatives). The score is standardized, ranging from from 0 to 100, with higher scores indicating a greater knowledge in docetaxel. Mean change in scores will be reported, as well as standard deviations.
Mean change in informed subscale of Decisional Conflict Scale over time | Up to 2 weeks
  The informed subscale of the Decisional Conflict Scale is comprised of 3 items given a score value of 0 = 'strongly agree to 4 = 'strongly disagree'. The items are summed, divided by 3, and then multiplied by 25. Scores range from 0 (feels extremely informed) to 100 (feels extremely uninformed).

SECONDARY OUTCOMES:
Proportion of invited participants who consent to the study | 1 day
  The proportion of participants who consented to the study from the total number of participants contacted will be reported.
Proportion of approached patients' providers who agree to be recorded | 1 day
  The proportion of approached patients' providers who agree to be recorded from the total number of patients' providers approached to participate will be reported.
Mean change in participant-reported anxiety over time | Up to 2 weeks
  The Patient-Reported Outcomes Measurement Information System (PROMIS) Anxiety Short form (4a) consists of 4 items addressing patient anxiety with item response scores ranging from 1 (never) to 5 (Always). Raw scores are converted to scaled T-scores with higher scores indicating a greater level of anxiety. Participants will be measured at baseline and 7 days post-appointment and compared over time.
Proportion of enrolled participants who create a recording | Up to 2 weeks
  The proportion of enrolled participants who created a recording of the total number of participants in the study will be reported.
Proportion of enrolled participants who listen to the recording | Up to 2 weeks
  The proportion of enrolled participants who listen to the recording or read its automatically generated transcript, measured by participant-reported survey at 7 days post-appointment of the total number of participants in the study will be reported.
Proportion of enrolled participants who report they received both mailed/emailed instructions to install/use the app | Up to 2 weeks
  The proportion of enrolled participants who report they received both mailed/emailed instructions to install/use the app measured by participant-reported survey at 7 days post-appointment of the total number of participants in the study will be reported.
Proportion of participants who report high shared decision-making effort | Up to 2 weeks
  High shared decision-making effort will be measured at 7 days post-appointment using the collaboRATE scale. The collaboRATE scale is a 3-item, 10-point Likert scale, where each encounter is scored as either '1' if the response to all three collaboRATE items is 9, or '0' if the response to any of the three collaboRATE items is less than 9. The percentage of all participants with a code of '1' will be calculated.
Proportion of patients who received docetaxel | Up to 30 days
  Docetaxel treatment received at 30 days post-appointment will be reported with a 95% confidence interval will be reported.
Proportion of patients who received docetaxel | Up to 60 days
  Docetaxel treatment received at 60 days post-appointment will be reported with a 95% confidence interval will be reported.

OTHER OUTCOMES:
Mean change in docetaxel knowledge score over time | Up to 28 days
  Change in docetaxel knowledge score is measured by participant report of knowledge using a docetaxel knowledge instrument, measured at baseline and 28 days post-appointment. The instrument was developed based on facts that patients and providers deem are important when making a treatment decision that includes docetaxel as an option for mCRPC (e.g., disease, prognosis, risks, benefits, alternatives). The score is standardized, ranging from from 0 to 100, with higher scores indicating a greater knowledge in docetaxel. Mean change in scores will be reported, as well as standard deviations.
Auto-generated transcript accuracy | Up to 60 days
  Auto-generated transcript accuracy will be measured by comparing the transcript to research staff transcription of the recording.
Quality of decision support and communication | Up to 60 days
  The Brief Decision Support Analysis Tool (DSAT-10) will be applied to recordings to evaluate treating physicians' and practitioners' use of decision support and communication skills with patients, with attention to docetaxel. Encounters are reviewed and scored on factors such as Decision making status, Knowledge of, Values/Preference associated with, Others' involvement with the decision, and Next Steps and given a score ranging from 1-10, with a higher score indicating a greater quality of decisional support.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Kwon, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kwon DH, Trihy L, Darvish N, Hearst E, Sumra S, Borno HT, Bose R, Chou J, de Kouchkovsky I, Desai A, Ekstrand B, Friedlander T, Kaur G, Koshkin VS, Nesheiwat S, Sepucha K, Small EJ, Aggarwal RR, Belkora J. Patients Can Administer Mobile Audio Recordings to Increase Knowledge in Advanced Prostate Cancer. Cancer Med. 2024 Nov;13(22):e70433. doi: 10.1002/cam4.70433. PMID 39569542